CLINICAL TRIAL: NCT07159555
Title: Neurofilaments Levels in Premature Newborns
Brief Title: Assessment of Neurofilaments Levels in Premature Newborns: Study of Their Early Development
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Collaborators: Centre Hospitalier Régional de la Citadelle (Other)
Responsible Party: Principal Investigator, Laurent Servais, Principal Investigator, Pediatrician, Centre Hospitalier Universitaire de Liege
Other Study IDs: Neurofilaments
Record Dates: First submitted 2025-08-28; First posted 2025-09-08 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Healthy Participants
Keywords: Healthy Participants; Neurofilament; Premature infant
MeSH Terms: conditions — Premature Birth | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neurofilament sampling in late preterm newborns: Late preterm infants (34-37 weeks of gestation) admitted to the neonatal unit. Up to 1 mL of additional blood will be collected during routine clinically indicated blood draws at birth, day 2, and weekly until 37 weeks of gestation. Samples will be analyzed for neurofilament concentrations. No independent venipuncture will be performed.
  Interventions: Other: Blood sampling for neurofilament analysis

INTERVENTIONS:
Other: Blood sampling for neurofilament analysis — An additional blood sample (maximum 1 mL) is collected during routine clinically indicated blood draws in late preterm infants (34-37 weeks of gestation). Samples are obtained at birth, day 2, and weekly until 37 weeks of gestation if blood draws are already planned. No separate venipuncture is performed. Samples are processed and stored for subsequent neurofilament concentration analysis.

SUMMARY:
This is a prospective observational study aiming to establish reference values of neurofilaments in late preterm newborns (34-37 weeks of gestation) and to evaluate their early postnatal evolution.

Neurofilaments are neuronal proteins released into the blood when nerve cells are damaged. They have emerged as promising biomarkers in neurodegenerative diseases, particularly in spinal muscular atrophy (SMA), where higher levels are associated with disease activity. However, very limited data exist on the normal dynamics of neurofilament levels in preterm infants.

In this study, up to 15 preterm newborns hospitalized in the neonatal unit will be enrolled (5 at 34 weeks, 5 at 35 weeks, 5 at 36 weeks of gestation). A maximum of 1 mL of additional blood will be collected only during routine clinically indicated blood draws, at birth, on day 2, and weekly until 37 weeks of gestation. Samples will be analyzed for neurofilament concentrations and compared across gestational ages, over time, and with existing data from term newborns and SMA patients.

The expected outcome is to generate normative data on neurofilament levels in late preterm infants, which will help interpret biomarker values in future studies and optimize early diagnosis and treatment strategies for neurodegenerative diseases such as SMA.

DETAILED DESCRIPTION:
Recent therapeutic advances in spinal muscular atrophy (SMA) have highlighted the importance of very early treatment, ideally before the onset of symptoms. Neurofilaments, structural proteins of neurons released into the blood when axons are damaged, have been identified as sensitive biomarkers of neurodegeneration and disease activity in SMA. Elevated neurofilament levels have been reported in affected infants, with a rapid decline following initiation of effective treatment.

Despite their growing importance as a biomarker, little is known about the normal postnatal dynamics of neurofilaments in preterm infants. Establishing normative data in this population is essential to correctly interpret biomarker levels in newborn screening programs and clinical follow-up, particularly for conditions such as SMA where treatment decisions rely on early biological signals.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 34 and 37 weeks of amenorrhea.
* Blood test scheduled for clinical reasons.
* Signed parental consent.

Exclusion Criteria:

* Known neurological disorders.
* Severe congenital malformations.
* Medical contraindication to blood sampling.

Max Age: 3 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Late preterm infants (34-37 weeks of gestation) admitted to the neonatal unit
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Neurofilament concentration in blood of late preterm infants | From birth to 37 weeks of gestational age (up to 3 weeks after inclusion depending on gestational age at birth).
  Measurement of blood neurofilament light chain (NfL) concentrations to establish reference values and describe their early postnatal evolution in late preterm infants.

SECONDARY OUTCOMES:
Postnatal evolution of neurofilament concentrations | From birth up to 37 weeks of gestational age (longitudinal follow-up).
  Analysis of changes in neurofilament levels over time in late preterm infants, from birth to 37 weeks of gestational age.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Servais, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Liege
Locations (1):
- Hopital Citadelle, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No